CLINICAL TRIAL: NCT04357977
Title: A Human Clinical Study to Collect Calibration and Performance Data for the RBA-2 Device
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kaligia Biosciences, LLC (Industry)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: KBS005
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus; COVID
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid +: Laboratory obtained Covid+ specimen results will be compared to saliva specimen
  Interventions: Diagnostic Test: RBA-2

INTERVENTIONS:
Diagnostic Test: RBA-2 — Collection of non-invasive in vivo saliva from confirmed cases of both infected and non-infected COVID-19 patients or site staff at the testing site and compare the test results using the RBA-2 against the standard test results used for diagnosis.

SUMMARY:
The current available diagnostic methods used for the detection of COVID-19 takes up to 4 hours. In some cases, these diagnostics tests make take up to a couple of days. As it is highly contagious, people who are in close contact with the infected person are at high risk of being infected. COVID-19 is transmitted through respiratory droplets produced when an infected person coughs or sneezes. The desire for rapid detection of COVID-19 has become an immediate necessity. The purpose of Kaligia Biosciences' saliva monitoring device (RBA-2) is to detect the presence of the COVID-19 virus in human saliva. The RBA-2 uses Raman Spectros-copy to detect the coronavirus. Once the sample is scanned successfully, the spectra contains the response of the component present in human saliva and provide results in a matter of minutes, rather than hours or days.

DETAILED DESCRIPTION:
The purpose of this study is to calibrate the performance of RBA-2 using people by comparing the results against a standard diagnostics test. The objective of this study is to collect non-invasive in vivo saliva from confirmed cases of both infected and non-infected COVID-19 patients or site staff at the testing site and compare the test results using the RBA-2 against the standard test results used for diagnosis.

The comparison of the results obtained from the current testing methods will be used to calibrate machine learning algorithms of the RBA-2.

ELIGIBILITY:
Inclusion Criteria:

Participants can be patients or staff members at the testing site.

Potential participants may be enrolled if:

1. They are identified as requiring a standard diagnostic test for COVID-19 or are being treated after testing positive for COVID-19;
2. They are age ≥ 18 years old;
3. They are willing and able to provide verbal informed consent.

Exclusion Criteria:

* Patients receiving active treatment with antivirals, chloroquine or immune modulators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients and study staff at the testing site who have been flagged for COVID-19 testing or who are being treated for COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Covid + | 10 days
  The comparison of the results obtained from the current testing methods will be used to calibrate machine learning algorithms of the RBA-2

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - AdventHealth Tampa, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Undecided